CLINICAL TRIAL: NCT01735617
Title: A Phase 2 Pilot Study to Characterize and Examine the Pharmacokinetics and Disease Bio-marker Response of Chronocort® in Adults With Congenital Adrenal Hyperplasia
Brief Title: Pilot Study to Characterize and Examine the Pharmacokinetics and Efficacy of Chronocort® in Adults With CAH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurocrine UK Limited (Industry)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DIUR-003
Record Dates: First submitted 2012-11-20; First posted 2012-11-28 (Estimated); Results first posted 2017-05-17 (Actual); Last update posted 2017-05-17 (Actual); Status verified 2017-04

CONDITIONS: Endocrine Disease; Adrenal Insufficiency; Congenital Adrenal Hyperplasia
Keywords: congenital adrenal hyperplasia; glucocorticoids; cortisol; adrenal
MeSH Terms: conditions — Endocrine System Diseases; Adrenal Insufficiency; Adrenal Hyperplasia, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hydrocortisone Modified Release Capsules (Experimental): Chronocort Modified Release Capsules, 5mg, 10mg and 20mg Dosing frequency twice-daily (mane and nocte) Dose setting by titration to achieve optimal biochemical and therapeutic response
  Interventions: Drug: Hydrocortisone Modified Release Capsules

INTERVENTIONS:
Drug: Hydrocortisone Modified Release Capsules — Patients with congenital adrenal hyperplasia standardised on conventional therapy is enrolled onto the study and treatment is switched to Chronocort, initially for pharmacokinetic assessment followed by longer-term biochemical and efficacy assessment
  Other Names: Chronocort

SUMMARY:
The purpose of this study is to gather safety and effectiveness information about a new formulation of Hydrocortisone (Chronocort®) used to treat patients with a disease called congenital adrenal hyperplasia (CAH). Hydrocortisone is the man-made version of the hormone cortisol, which is released in the body following a regular daily pattern. The objective of the study is to measure the levels of hydrocortisone that are absorbed into the bloodstream once Chronocort® is taken and what affects it has on other hormones in the body. Since Chronocort® is anticipated to mimic the same release pattern of cortisol in the body, it is hoped that patients with CAH will be treated more effectively to manage their disease.

DETAILED DESCRIPTION:
This study is a Phase 2 pilot study to characterize and examine the pharmacokinetics and efficacy profile of Chronocort® in adults with congenital adrenal hyperplasia (CAH). It is designed as a two-part, single cohort, open label, multiple dose Phase 2 pilot study to: (Part A) characterize and examine the pharmacokinetics (PK) and disease bio-marker behavior following short-term dosing with Chronocort®; and to (Part B) examine the disease control after six months dose titration with Chronocort® in adults with CAH.

ELIGIBILITY:
Inclusion Criteria:

1. Known CAH due to 21-hydroxylase deficiency (classic CAH) based on hormonal and genetic testing currently treated with hydrocortisone, prednisone, prednisolone or dexamethasone on a stable dosage for a minimum of 3 months.
2. Male or female patients aged 18 and above.
3. Provision of signed written informed consent.
4. Good general health.
5. Females of childbearing potential must have a negative pregnancy test initially and at all visits. Females who are engaging in sexual intercourse must be using a medically acceptable method of contraception (as defined in the protocol, section 10.5).
6. Plasma renin activity must be within the clinically acceptable range at screening (less than 1.5 times upper normal range).

Exclusion Criteria:

1. Co-morbid condition requiring daily administration of a medication that induces hepatic enzymes or interferes with the metabolism of glucocorticoids.
2. Clinical or biochemical evidence of hepatic or renal disease. Creatinine above the normal range or elevated liver function tests (ALT or AST) > 2 times the upper limits of normal.
3. Females who are pregnant or lactating.
4. Women taking an estrogen-containing oral contraceptive pill and who have taken it within 6 weeks of recruitment.
5. Patients taking spironolactone.
6. Patients on inhaled or oral steroids apart from treatment for CAH.
7. Patients with any other significant medical or psychiatric conditions that in the opinion of the Investigator would preclude participation in the trial.
8. Participation in another clinical trial of an investigational or licensed drug or device within the 3 months prior to inclusion in this study.
9. Patients with history of bilateral adrenalectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah P Merke, BS, MS, MD, Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mallappa A, Sinaii N, Kumar P, Whitaker MJ, Daley LA, Digweed D, Eckland DJ, Van Ryzin C, Nieman LK, Arlt W, Ross RJ, Merke DP. A phase 2 study of Chronocort, a modified-release formulation of hydrocortisone, in the treatment of adults with classic congenital adrenal hyperplasia. J Clin Endocrinol Metab. 2015 Mar;100(3):1137-45. doi: 10.1210/jc.2014-3809. Epub 2014 Dec 11. PMID 25494662

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydrocortisone Modified Release Capsules
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All treated subjects
Arm/Group | Hydrocortisone Modified Release Capsules
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.7 (12.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 13
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic Profile (Cmax) Following Short-term Treatment With Chronocort® in Adult Patients With Congenital Adrenal Hyperplasia
Description: The maximum plasma concentration (Cmax) of chronocort
Time Frame: 24 hours
Population: All treated subjects
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Chronocort: Chronocort Modified Release Capsules 10 mg twice-daily.
Arm/Group | Chronocort
Number analyzed (Participants) | 16
nmol/L | 601.213 (114.5987)
Statistical Analysis 1: Comparison: Chronocort; The pharmacokinetic profile was characterised by an overnight rise in cortisol levels reaching a maximal concentration approximately 8 hours post dosing; Test type: Superiority or Other; Geometric means = 563.38, Standard Deviation 162.51

2. Primary Outcome: Pharmacokinetic Profile (AUC0-24) Following Short-term Treatment With Chronocort® in Adult Patients With Congenital Adrenal Hyperplasia
Description: Area under the curve (AUC) from 0 to 24 hours (sampling occurs at the following timepoints: 2300, 0100, 0300, 0500, 0600, 0700, 0800, 0900, 1000, 1100, 1200, 1300, 1400, 1500, 1600, 1700, 1900, 2100, 2300hrs)
Time Frame: 24 hours (at 2300, 0100, 0300, 0500, 0600, 0700, 0800, 0900, 1000, 1100, 1200, 1300, 1400, 1500, 1600, 1700, 1900, 2100, 2300hrs)
Population: All treated subjects
Measure: Mean (Standard Deviation); unit: h*nmol/L
Groups:
- Chroncort: Chronocort Modified Release Capsules 10mg twice-daily
Arm/Group | Chroncort
Number analyzed (Participants) | 16
h*nmol/L | 5027.641 (1247.8425)

3. Primary Outcome: Pharmacokinetic Profile (Tmax) Following Short-term Treatment With Chronocort® in Adult Patients With Congenital Adrenal Hyperplasia
Description: Time to maximum plasma concentration (tmax)
Time Frame: 24 hours
Population: All treated subjects
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Chronocort: Chronocort Modified Release Capsules 10mg twice-daily
Arm/Group | Chronocort
Number analyzed (Participants) | 16
Hours | 7.9 (2.9)

4. Secondary Outcome: The Percentage of Patients With 17-OHP and Androstenedione Levels at 0700h Within Proposed Optimal Ranges Whilst on Chronocort and Whilst on Standard Therapy (at Baseline)
Description: Proposed optimal ranges of 17-OHP: 300-1200ng/dl Proposed optimal ranges of androstenedione: 40-150ng.dl for males and 30-200ng/dl for females
Time Frame: Specific time point (0700hrs)
Measure: Number; unit: percentage of participants
Arm/Group | Hydrocortisone Modified Release Capsules
Number analyzed (Participants) | 16
percentage of participants
  17-OHP (baseline) | 0
  17-OHP (final visit) | 12.5
  Androstenedione (baseline) | 56.3
  Androstenedione (final visit) | 81.3

5. Secondary Outcome: 17-OHP Levels at 0700h, 1700h and 2300h
Description: 17-OHP levels at 0700h, 1700h and 2300h
Time Frame: Specified time points (0700h, 1700h and 2300h)
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Hydrocortisone Modified Release Capsules
Number analyzed (Participants) | 16
nmol/L
  17-OHP: Part A, Days 1-2 (0700h) | 76.97 (91.986)
  17-OHP: Part A, Days 1-2 (1700h) | 70.99 (104.106)
  17-OHP: Part A, Days 1-2 (2300h) | 55.35 (93.632)
  17-OHP: Part A, Days 4-5 (0700h) | 7.72 (8.231)
  17-OHP: Part A, Days 4-5 (1700h) | 23.55 (66.046)
  17-OHP: Part A, Days 4-5 (2300h) | 27.27 (55.140)
  17-OHP: Part B, Visit 2 (0700h) | 24.86 (54.086)
  17-OHP: Part B, Visit 2 (1700h) | 15.17 (20.400)
  17-OHP: Part B, Visit 2 (2300h) | 26.65 (51.185)
  17-OHP: Part B, Visit 3 (0700h) | 34.87 (49.072)
  17-OHP: Part B, Visit 3 (1700h) | 13.81 (20.700)
  17-OHP: Part B, Visit 3 (2300h) | 18.95 (28.276)
  17-OHP: Part B, Visit 4 (0700h) | 13.67 (19.091)
  17-OHP: Part B, Visit 4 (1700h) | 34.70 (69.876)
  17-OHP: Part B, Visit 4 (2300h) | 22.19 (46.826)

6. Secondary Outcome: Androstenedione Levels at 0700h, 1700h and 2300h
Description: Androstenedione levels at 0700h, 1700h and 2300h
Time Frame: Specified time points (0700h, 1700h and 2300h)
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Hydrocortisone Modified Release Capsules
Number analyzed (Participants) | 16
nmol/L
  Androstenedione: Part A, Days 1-2 (0700h) | 7.92 (8.474)
  Androstenedione: Part A, Days 1-2 (1700h) | 7.54 (7.966)
  Androstenedione: Part A, Days 1-2 (2300h) | 7.43 (9.388)
  Androstenedione: Part A, Days 4-5 (0700h) | 3.11 (2.178)
  Androstenedione: Part A, Days 4-5 (1700h) | 4.62 (8.005)
  Androstenedione: Part A, Days 4-5 (2300h) | 5.37 (8.340)
  Androstenedione: Part B, Visit 2 (0700h) | 4.96 (6.731)
  Androstenedione: Part B, Visit 2 (1700h) | 3.47 (3.094)
  Androstenedione: Part B, Visit 2 (2300h) | 3.79 (3.748)
  Androstenedione: Part B, Visit 3 (0700h) | 4.57 (3.561)
  Androstenedione: Part B, Visit 3 (1700h) | 3.61 (2.713)
  Androstenedione: Part B, Visit 3 (2300h) | 3.91 (3.103)
  Androstenedione: Part B, Visit 4 (0700h) | 3.40 (1.973)
  Androstenedione: Part B, Visit 4 (1700h) | 4.19 (4.602)
  Androstenedione: Part B, Visit 4 (2300h) | 3.37 (2.655)

7. Secondary Outcome: ACTH Levels at 0700h, 1700h and 2300h
Description: ACTH levels at 0700h, 1700h and 2300h
Time Frame: Specified time points (0700h, 1700h and 2300h)
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Hydrocortisone Modified Release Capsules
Number analyzed (Participants) | 16
pmol/L
  ACTH: Part A, Days 1-2 (0700h) | 21.06 (29.767)
  ACTH: Part A, Days 1-2 (1700h) | 20.93 (30.121)
  ACTH: Part A, Days 1-2 (2300h) | 7.75 (9.873)
  ACTH: Part A, Days 4-5 (0700h) | 4.16 (9.190)
  ACTH: Part A, Days 4-5 (1700h) | 4.71 (7.382)
  ACTH: Part A, Days 4-5 (2300h) | 7.37 (7.990)
  ACTH: Part B, Visit 2 (0700h) | 7.02 (12.159)
  ACTH: Part B, Visit 2 (1700h) | 5.57 (6.769)
  ACTH: Part B, Visit 2 (2300h) | 8.66 (14.637)
  ACTH: Part B, Visit 3 (0700h) | 9.66 (12.418)
  ACTH: Part B, Visit 3 (1700h) | 4.71 (6.331)
  ACTH: Part B, Visit 3 (2300h) | 6.04 (7.997)
  ACTH: Part B, Visit 4 (0700h) | 12.18 (29.911)
  ACTH: Part B, Visit 4 (1700h) | 13.66 (22.851)
  ACTH: Part B, Visit 4 (2300h) | 9.44 (17.474)

8. Secondary Outcome: AUC Values (Nmol*h/L) for Androstenedione
Description: AUC values (nmol*h/L) for Androstenedione for the following reporting periods: 24 hours (2300-2300h), 2300-0700h, 0700-1500h and 1500-2300h
Time Frame: Specific time points (2300-2300h, 2300-0700h, 0700-1500h and 1500-2300h)
Measure: Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | Hydrocortisone Modified Release Capsules
Number analyzed (Participants) | 16
nmol*h/L
  Androstenedione: Part A, Days 1-2 AUC (2300-2300h) | 166.19 (171.969)
  Androstenedione: Part A, Days 1-2 AUC (2300-0700h) | 41.42 (34.133)
  Androstenedione: Part A, Days 1-2 AUC (0700-1500h) | 65.33 (76.337)
  Androstenedione: Part A, Days 1-2 AUC (1500-2300h) | 59.44 (65.995)
  Androstenedione: Part A, Days 4-5 AUC (2300-2300h) | 104.37 (128.725)
  Androstenedione: Part A, Days 4-5 AUC (2300-0700h) | 36.02 (40.225)
  Androstenedione: Part A, Days 4-5 AUC (0700-1500h) | 32.01 (31.503)
  Androstenedione: Part A, Days 4-5 AUC (1500-2300h) | 37.91 (58.394)
  Androstenedione: Part B, Visit 2 AUC (2300-2300h) | 88.58 (86.364)
  Androstenedione: Part B, Visit 2 AUC (2300-0700h) | 35.12 (43.580)
  Androstenedione: Part B, Visit 2 AUC (0700-1500h) | 26.07 (22.298)
  Androstenedione: Part B, Visit 2 AUC (1500-2300h) | 27.39 (23.989)
  Androstenedione: Part B, Visit 3 AUC (2300-2300h) | 91.46 (65.295)
  Androstenedione: Part B, Visit 3 AUC (2300-0700h) | 33.25 (26.255)
  Androstenedione: Part B, Visit 3 AUC (0700-1500h) | 27.92 (16.297)
  Androstenedione: Part B, Visit 3 AUC (1500-2300h) | 30.30 (26.188)
  Androstenedione: Part B, Visit 4 AUC (2300-2300h) | 86.27 (70.892)
  Androstenedione: Part B, Visit 4 AUC (2300-0700h) | 29.09 (23.314)
  Androstenedione: Part B, Visit 4 AUC (0700-1500h) | 27.03 (20.009)
  Androstenedione: Part B, Visit 4 AUC (1500-2300h) | 30.13 (28.797)

9. Secondary Outcome: AUC Values (Nmol*h/L) for 17-OHP
Description: AUC values (nmol*h/L) for 17-OHP for the following reporting periods: 24 hours (2300-2300h), 2300-0700h, 0700-1500h and 1500-2300h
Time Frame: Specific time points (2300-2300h, 2300-0700h, 0700-1500h and 1500-2300h)
Measure: Mean (Standard Deviation); unit: nmol*h/L
Arm/Group | Hydrocortisone Modified Release Capsules
Number analyzed (Participants) | 16
nmol*h/L
  17-OHP: Part A, Days 1-2 AUC 2300-2300h | 1407.83 (1829.291)
  17-OHP: Part A, Days 1-2 AUC 2300-0700h | 243.99 (339.580)
  17-OHP: Part A, Days 1-2 AUC 0700-1500h | 607.74 (805.822)
  17-OHP: Part A, Days 1-2 AUC 1500-2300h | 556.11 (769.492)
  17-OHP: Part A, Days 4-5 AUC 2300-2300h | 446.90 (817.074)
  17-OHP: Part A, Days 4-5 AUC 2300-0700h | 169.83 (268.178)
  17-OHP: Part A, Days 4-5 AUC 0700-1500h | 91.53 (147.801)
  17-OHP: Part A, Days 4-5 AUC 1500-2300h | 190.73 (425.505)
  17-OHP: Part B, Visit 2 AUC 2300-2300h | 395.65 (587.533)
  17-OHP: Part B, Visit 2 AUC 2300-0700h | 168.01 (337.666)
  17-OHP: Part B, Visit 2 AUC 0700-1500h | 82.41 (91.708)
  17-OHP: Part B, Visit 2 AUC 1500-2300h | 145.24 (215.115)
  17-OHP: Part B, Visit 3 AUC 2300-2300h | 432.02 (393.897)
  17-OHP: Part B, Visit 3 AUC 2300-0700h | 152.63 (144.576)
  17-OHP: Part B, Visit 3 AUC 0700-1500h | 139.21 (147.353)
  17-OHP: Part B, Visit 3 AUC 1500-2300h | 140.18 (182.786)
  17-OHP: Part B, Visit 4 AUC 2300-2300h | 436.54 (678.052)
  17-OHP: Part B, Visit 4 AUC 2300-0700h | 101.33 (148.003)
  17-OHP: Part B, Visit 4 AUC 0700-1500h | 120.32 (172.134)
  17-OHP: Part B, Visit 4 AUC 1500-2300h | 214.89 (364.641)

10. Secondary Outcome: AUC Values (Pmol*h/L) for ACTH
Description: AUC values (pmol*h/L) for ACTH for the following reporting periods: 24 hours (2300-2300h), 2300-0700h, 0700-1500h and 1500-2300h
Time Frame: Specific time points (2300-2300h, 2300-0700h, 0700-1500h and 1500-2300h)
Measure: Mean (Standard Deviation); unit: pmol*h/L
Arm/Group | Hydrocortisone Modified Release Capsules
Number analyzed (Participants) | 16
pmol*h/L
  ACTH: Part A, Days 1-2 AUC (2300-2300h) | 356.25 (415.949)
  ACTH: Part A, Days 1-2 AUC (2300-0700h) | 54.72 (70.267)
  ACTH: Part A, Days 1-2 AUC (0700-1500h) | 166.18 (206.294)
  ACTH: Part A, Days 1-2 AUC (1500-2300h) | 135.35 (169.002)
  ACTH: Part A, Days 4-5 AUC (2300-2300h) | 120.00 (121.454)
  ACTH: Part A, Days 4-5 AUC (2300-0700h) | 52.22 (62.067)
  ACTH: Part A, Days 4-5 AUC (0700-1500h) | 21.29 (19.824)
  ACTH: Part A, Days 4-5 AUC (1500-2300h) | 47.13 (57.145)
  ACTH: Part B, Visit 2 AUC (2300-2300h) | 125.45 (118.081)
  ACTH: Part B, Visit 2 AUC (2300-0700h) | 43.09 (46.711)
  ACTH: Part B, Visit 2 AUC (0700-1500h) | 34.14 (48.423)
  ACTH: Part B, Visit 2 AUC (1500-2300h) | 48.22 (49.078)
  ACTH: Part B, Visit 3 AUC (2300-2300h) | 154.10 (172.474)
  ACTH: Part B, Visit 3 AUC (2300-0700h) | 50.02 (57.268)
  ACTH: Part B, Visit 3 AUC (0700-1500h) | 52.46 (64.571)
  ACTH: Part B, Visit 3 AUC (1500-2300h) | 51.63 (70.735)
  ACTH: Part B, Visit 4 AUC (2300-2300h) | 252.30 (420.220)
  ACTH: Part B, Visit 4 AUC (2300-0700h) | 58.80 (107.955)
  ACTH: Part B, Visit 4 AUC (0700-1500h) | 110.58 (329.386)
  ACTH: Part B, Visit 4 AUC (1500-2300h) | 82.92 (120.287)

ADVERSE EVENTS:
Time Frame: Approximately 7 months
Arm/Group | Hydrocortisone Modified Release Capsules
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 16/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydrocortisone Modified Release Capsules (N=16)
Headache (Nervous system disorders) | 13 (13)
Fatigue (General disorders) | 13 (13)
Anaemia (Blood and lymphatic system disorders) | 7 (9)
Dizziness (Nervous system disorders) | 8 (8)
Weight increase (Investigations) | 7 (7)
Appetite decrease (Metabolism and nutrition disorders) | 7 (7)
Appetite increase (Metabolism and nutrition disorders) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 5 (5)
Acne (Skin and subcutaneous tissue disorders) | 5 (5)
Asthenia (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No